CLINICAL TRIAL: NCT06991335
Title: Deep Brain Stimulation (DBS) of the Ventral Capsule Ventral Striatum (VC/VS) for the Treatment of Apathy in Parkinson's Disease (PD)
Brief Title: VC/VS for Apathy in PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nora Vanegas (Other)
Responsible Party: Sponsor-Investigator, Nora Vanegas, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-57525
Record Dates: First submitted 2025-05-20; First posted 2025-05-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Deep Brain Stimulation; Apathy
Keywords: parkinson disease; deep brain stimulation; apathy; dbs; pd; neuromodulation; imaging
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Medtronic Percept PC with SenSight Directional Leads will be implanted to control the shape and size of stimulation

SUMMARY:
Apathy is a disabling neuropsychiatric symptom marked by reduced goal-directed behavior, including diminished interest, motivation, emotional expression, and social engagement. Though not formally defined in the DSM-V, apathy is common in several neurological and psychiatric disorders and significantly affects quality of life. In Parkinson's Disease (PD), it affects about 40% of patients and is associated with increased caregiver burden, reduced functional ability, and nearly threefold higher mortality.

PD affects over 680,000 Americans today and is projected to impact more than 1.2 million by 2030. It presents with both motor symptoms (e.g., bradykinesia, tremor, rigidity) and non-motor symptoms like depression, anxiety, and apathy. While motor symptoms are often managed with dopaminergic medications and deep brain stimulation (DBS) targeting motor regions (e.g., subthalamic nucleus, globus pallidus internal), apathy typically persists or worsens following these treatments. No FDA-approved or consistently effective treatments exist for apathy in PD. Dopamine agonists may help but have side effects that limit long-term use. SSRIs and cholinesterase inhibitors may be tried for co-occurring depression or cognitive decline, but they are not indicated for apathy and can worsen symptoms or cause adverse effects in PD.

This protocol proposes targeting apathy in PD using DBS of the ventral capsule/ventral striatum (VC/VS), a region involved in reward processing and goal-directed behavior. VC/VS DBS is FDA-approved under a Humanitarian Device Exemption for OCD and has shown promise in treating depression, addiction, and other disorders involving motivational deficits. Neuroimaging and preclinical models strongly implicate this region in the regulation of goal-directed behavior, reward sensitivity, and cognitive control-mechanisms disrupted in apathy. Stimulating VC/VS may improve motivation through fibers connected to orbitofrontal and anterior cingulate cortices (reward sensitivity) and dorsal prefrontal regions (cognitive control).

Support for this approach comes from a case report where a patient with PD and OCD received both STN and VC/VS DBS. In addition to motor and OCD symptom improvement, the patient showed a significant reduction in apathy. Apathy worsened when stimulation ceased and improved again when resumed, suggesting a causal relationship. VC/VS DBS was safe, did not impair motor symptoms, and appeared to enhance motivation.

This study aims to test the safety and efficacy of VC/VS DBS for apathy in PD. Building on extensive animal, imaging, and clinical data, it addresses a major unmet need using an existing DBS platform. The approach is supported by established neurocircuitry, prior clinical experience with VC/VS targeting, and early evidence suggesting potential benefit. It does not duplicate prior studies but extends DBS to a new, underserved indication within PD.

DETAILED DESCRIPTION:
Apathy is a significant mental health condition. Apathy was originally defined as a disorder of motivation and is now operationalized as a reduction in goal-directed behavior. It manifests with diminished interest, goal setting, emotional expression, and social connection. Although not named as a formal diagnosis in the DSM-V, apathy is highly prevalent and co-morbid with several neuropsychiatric disorders. Apathy impacts ~40% of patients with Parkinson's Disease (PD), ~60% of patients with Alzheimer's Disease, ~40% of patients with major depressive disorder, ~50% of patients with schizophrenia and more than 30% of individuals after stroke. Its presence conveys greater caregiver burden, poorer engagement in activities of daily living, higher risk of cognitive decline, and generally lower quality of life. These factors impose a profound clinical, social, and economic burden, not only by exacerbating the challenges faced by individuals with apathy but also by straining caregivers, healthcare, and societal resources.

In the US alone, PD impacts over 680,000 individuals today and is anticipated to impact 1,238,000 individuals by 2030. PD is a neuropsychiatric disorder characterized by a combination of motor symptoms including bradykinesia (100%), tremor (70-90%), and rigidity (90%) and non-motor symptoms, including psychiatric issues such as depression (50%), anxiety (40%) and apathy (40%). Apathy is now recognized as one of the most debilitating nonmotor symptoms. It is associated with decreased participation in everyday activities, decreased functional capabilities, and increased caregiver burden. Remarkably, apathetic PD patients have a nearly 3X increased risk of mortality compared to their non-apathetic counterparts.

Dopaminergic medications and deep brain stimulation (DBS) of the subthalamic nucleus (STN) or the globus pallidus internus (GPi) are effective treatments for the motor complications of PD. However, apathy symptoms commonly persist and may even worsen after DBS, with most patients continuing to deteriorate over time with significant implications on their quality of life and overall morbidity and mortality. Furthermore, although dopamine agonists (e.g., Pramipexole, Ropinirole, Rotigotine), may reduce apathy severity in PD, they commonly lead to side effects including psychosis and impulse control disorders that limit their prolonged use. Therefore, there are no effective and practically usable treatments for apathy in PD. Importantly, other neuropsychiatric symptoms such as depression and cognitive decline often co-occur in PD patients with apathy. In cases of co-morbid depression, apathy may be clinically distinguished, and treatment options for depression may be attempted (e.g., selective serotonin reuptake inhibitors, SSRIs). However, the use of SSRI antidepressants has been associated with greater apathy in PD and are not indicated specifically for the treatment of apathy. Similarly, cholinesterase inhibitors (e.g., rivastigmine, galantamine) may be attempted in patients with apathy and associated cognitive impairment. However, common side effects (i.e., psychosis, confusion, anxiety) are frequently prohibitive in PD and limit their use. Thus, in light of the lack of specific treatments for apathy in PD, the detrimental impact of apathy on quality of life, morbidity, and mortality in PD represents a critical treatment gap.

The success of DBS for the treatment of motor symptoms in PD derives from the well understood pathophysiology within the underlying circuit. Analogously, the investigators propose to leverage our understanding of the circuitry underlying apathy as a disruption of goal-directed behavior to rationally target the treatment of apathy. In humans, tasks studying goal-directed behavior consistently implicate the region of the ventral striatum (VS) and adjacent white matter of the ventral portion of the anterior limb of the internal capsule (ventral capsule, VC), which carries axons from prefrontal cortex (PFC). DBS of this region is used to treat refractory OCD (under US FDA humanitarian device exemption status), as well as depression, addiction, and other disorders (as investigational indications). The emerging success of neuromodulation of this region for such a diversity of disorders strongly suggests common underlying mechanisms. Two prominent mechanisms likely playing important roles are reward sensitivity and cognitive control. Deficits in reward sensitivity may manifest as anhedonia or avoidance, and deficits in cognitive control may produce inattention or effort intolerance. Aspects of these deficits appear in various combinations in OCD, depression, addiction, and other disorders treated by VC/VS DBS. Stimulation in this region likely enhances reward sensitivity via fibers from the orbitofrontal and ventral anterior cingulate cortices and the VS and likely exerts influence on cognitive control via stimulation of fibers from dorsal PFC and the dorsal anterior cingulate cortex. Deficits in goal-directed behavior may be attributable to either/both of these dimensions of dysfunction, motivating our hypothesis that VC/VS of this region will ameliorate apathy.

Indeed, further evidence for this therapeutic strategy comes from a case report in which a single patient was implanted bilaterally in both the STN and VC/VS for treatment of motor symptoms in PD and treatment-resistant OCD, respectively. In addition to achieving improvement in motor and OCD symptoms, VC/VS DBS also led to a significant reduction in apathy severity. During an unplanned discontinuation of stimulation due to battery depletion, OCD symptoms and apathy abruptly worsened. When VC/VS stimulation resumed, OCD and apathy once again improved. Even though this is a single case study, it suggests that 1) a dual implant (VC/VS + motor target) is safe and tolerable in PD; 2) VC/VS DBS in PD does not worsen motor symptoms; 3) VC/VS DBS shows promise for improving apathy in PD.

This protocol aims to address apathy/loss of motivation, one of the most disabling and largely undertreated symptoms of PD, with VC/VS DBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disorder as defined by the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease (MDS-PD).
* Presence of severe apathy as determined by apathy criteria established by the International Society for Central Nervous System Clinical Trials and Methodology Apathy Working Group (ISCTM-AWG).
* Apathy severity of -9 to +36, on the Lille Apathy Rating Scale (LARS) for at least 2 years.
* Documentation by primary neurologist of refractoriness to treatment for apathy with at least two dopamine-based treatments (e.g., levodopa, dopamine agonist) of sufficient dose and duration.
* Pre-DBS neuropsychological testing indicating normal cognition. Participants with mild cognitive impairment who have been evaluated by a cognitive neurologist for consideration of treatment (i.e., cholinesterase inhibitor) if indicated, may be included in the study once treatment has been stabilized for at least 2 months.
* Ability and willingness to give informed consent.
* Presence of a caregiver/informant who can complete study surveys/interviews related to the study participant.
* Stability of antidepressant medication dosing (i.e., SSRIs, Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs), etc.) for a minimum of four weeks prior to surgery.

Exclusion Criteria:

* Major neurocognitive disorder (i.e., dementia) as determined by pre-DBS neuropsychological testing.
* Explanation of apathy symptoms by comorbid depression as determined by a psychiatric interview including the Montgomery and Asberg depression rating scale (MADRS). Individuals with a MADRS score ≥15 will be excluded.
* History of suicide attempt in the past 36 months or current active suicidal ideation (Yes to #2-5 on the Columbia Suicide Severity Rating Scale - C-SSRS).
* Current PD-related psychosis (e.g., visual hallucinations).
* Any psychiatric, neurological and/or medical condition that makes the subject, in the opinion of the investigators, a poor candidate.
* Alcohol/substance use disorder, moderate or severe, within the previous 12 months.
* Female who is pregnant or breastfeeding or has plans to become pregnant in the next 24 months.
* Any contraindication for MRI.
* Presence of any of the following disorders: a) central nervous system infection, b) toxic-metabolic encephalopathy, defined as a syndrome of delirium associated with an identifiable toxin such as a chemical or metabolic disorder, c) multiple sclerosis, d) developmental delay.
* Need for diathermy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2032-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Apathy Symptoms | 9 to 15 months
  Response will be defined as a reduction of ≥3 points on the Apathy Evaluation Scale (AES) and Clinical Global Impression Scale - Improvement (CGI-I) of 1 or 2 (indicating 1=very much improved or 2=much improved). Higher AES scores are associated with higher apathy levels. Lower CGI-I scores indicate greater improvement in the participant's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Vanegas-Arroyave, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code